CLINICAL TRIAL: NCT06152458
Title: Blessing or Curse? Combined Vitamin Therapy in Non Viral Septic Shock.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7849-PTE 2019
Record Dates: First submitted 2023-09-01; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Septic Shock
Keywords: sepsis; vitamin-c; thiamine; septic shock
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Ascorbic Acid; Thiamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Patients in the intervention group (n=23) received the combined vitamin therapy: IV vitamin C (1.5 g every 6 hours administered as an infusion over 30 to 60 minutes and mixed in a 100- mL solution of normal saline), hydrocortisone (100 mg in bolus-100 mg in perfusor up to 60 min (200mg 24h),), and thiamine (200 mg every 12 hours administered as an infusion over 30 to 60 minutes and mixed in a 100-mL solution of normal saline) for 3 days.
  Interventions: Drug: Vitamin C
- control group (No Intervention): As a control group, we selected 20 age- and sex-matched patients with septic shock who did not receive vitamin treatment.They received the standard of care for septic shock.

INTERVENTIONS:
Drug: Vitamin C — Patients in the intervention group (G1) (n=23) received the combined vitamin therapy: IV vitamin C (1.5 g every 6 hours administered as an infusion over 30 to 60 minutes and mixed in a 100- mL solution of normal saline), hydrocortisone (100 mg in bolus-100 mg in perfusor up to 60 min (200mg 24h),), and thiamine (200 mg every 12 hours administered as an infusion over 30 to 60 minutes and mixed in a 100-mL solution of normal saline) for 3 days.
  Other Names: Thiamine
  Arms: intervention group

SUMMARY:
Introduction: Septic shock leads to high morbidity and mortality in critically ill patients. Several lower-case scientific studies have supported the synergistic positive effect of vitamin C, thiamine, and hydrocortisone on sepsis-induced organ dysfunction.

Aim: Our aim was to investigate the effect of vitamin complex on organ failure, laboratory parameters, respiratory and antibiotic treatment, intensive care time, and mortality in septic shock patients.

Material and methods: In our retrospective and prospective analysis, we collected parameters from 43 (23 vitamin-treated, 20 control) septic shock patients. Patients treated with vitamin, they received vitamin C (4x1500 mg), thiamine (2x200 mg) for three days (2). In other respects, and for hydrocortisone (200 mg / 24h), both groups of patients received treatment according to the European Sepsis Recommendation. SPSS (V-21) data were used for data collection, Kolmogorov-Smirnov, Wilcoxon, Mann-Whitney U tests were used for statistical analysis.

Ethical license: 7849-PTE 2019.

ELIGIBILITY:
Inclusion Criteria:

* septic shock
* intensive care unit administration

Exclusion Criteria:

* under age 18
* above age 80
* moribund patients
* pregnant patients
* active kidney stone
* inability to obtain consent
* viral or mixed sepsis
* missed dose of vitamin C/ thiamin or hydrocortisone
* Physician refused
* Vitamin C / Thiamine/ Hydrocortisone for other indications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
ventilation | intensive care unit discharge (up to 90 days)
  duration of mechanical ventilation (days)
vasopressors | intensive care unit discharge (up to 90 days)
  length of circulatory support (days)
Length of stay | intensive care unit discharge (up to 90 days)
  length of Intensive care unit staying (days)
main mortality | intensive care unit discharge (up to 90 days)
  all-cause mortality (dead/survived) in the intensive care unit

SECONDARY OUTCOMES:
secondary outcomes | up to 5 days after admission to intensive care
  development of inflammatory laboratory parameters:
  - se-carbamide (mg/dl)
secondary outcomes | up to 5 days after admission to intensive care
  development of inflammatory laboratory parameters:
  - se-creatinine (µmol/L)
secondary outcomes | up to 5 days after admission to intensive care
  development of inflammatory laboratory parameters:
  - plateletes (G/L),
secondary outcomes | up to 5 days after admission to intensive care
  development of inflammatory laboratory parameters:
  - procalcitonin (ng/ml),
secondary outcomes | up to 5 days after admission to intensive care
  development of inflammatory laboratory parameters:
  - white blood cells (G/L)
secondary outcomes | up to 5 days after admission to intensive care
  development of inflammatory laboratory parameters:
  - heat shock C-reactive protein (mg/L)
secondary outcomes | up to 5 days after admission to intensive care
  development of inflammatory laboratory parameters:
  - se-lactate (mmol/L)
antibiotics | intensive care unit discharge (up to 90 days)
  the length of antibiotic treatment (days)
PiCCO parameters | up to 5 days after admission to intensive care
  changes in invasive hemodynamic parameters-PiCCO ®:
  - cardiac index (l/min/m2)
PiCCO parameters | up to 5 days after admission to intensive care
  changes in invasive hemodynamic parameters-PiCCO ®:
  - extravascular lung water (ml/kg)
PiCCO parameters | up to 5 days after admission to intensive care
  changes in invasive hemodynamic parameters-PiCCO ®:
  - intrathoracic body water (ml/m2)
PiCCO parameters | up to 5 days after admission to intensive care
  changes in invasive hemodynamic parameters-PiCCO ®:
  - myocardial contractility (dP/dTmax- (mm hg/s)
other mortality's | up to 60 days after admission to intensive care
  in-hospital, 30- and 60-day mortality (dead/survived)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesia and Intensive Therapy University of Pecs, Pécs, Baranya, Hungary